Early diagnosis of anastomotic leakage after colorectal surgery: a prospective observational validation study of the Dutch Leakage score, serum procalcitonin and serum CRP: the Italian ColoRectal Anastomotic Leakage (iCRAL) study group.

#### **BACKGROUND**

Anastomotic leakage is a dreaded major complication after colorectal surgery [1]. The overall incidence of anastomotic dehiscence and subsequent leaks is 2 to 7 percent when performed by experienced surgeons [2-5]. The lowest leak rates are found with ileocolic anastomoses (1 to 3 percent) and the highest occur with coloanal anastomosis (10 to 20 percent) [6]. Leaks usually become apparent between five and seven days postoperatively. Almost half of all leaks occur after the patient has been discharged, and up to 12 percent occur after postoperative day 30 [4]. Late leaks often present insidiously with low-grade fever, prolonged ileus, and nonspecific symptoms attributable to other postoperative infectious complications. Small, contained leaks present later in the clinical course and may be difficult to distinguish from postoperative abscesses by radiologic imaging, making the diagnosis uncertain and underreported.

There is no uniform definition of an anastomotic dehiscence and leak [5]. In a review of 97 studies, as an example, 56 different definitions of an anastomotic leak were used [7]. The majority of reports define an anastomotic leak using clinical signs, radiographic findings, and intraoperative findings [8, 9]. The clinical signs include: Pain, Fever, Tachycardia, Peritonitis, Feculent drainage, Purulent drainage. The radiographic signs include: Fluid collections, Gas containing collections. The intraoperative findings include: Gross enteric spillage, Anastomotic disruption.

Risk factors for a dehiscence and leak are classified according to the site of the anastomosis (extraperitoneal or intraperitoneal). A prospective review of 1598 patients undergoing 1639 anastomotic procedures for benign or malignant colorectal disease found a significantly increased ALL 3 – Protocollo dello Studio

risk of anastomotic leak with extraperitoneal compared with intraperitoneal anastomoses (6.6 versus 1.5 percent; 2.4 percent overall) [10].

Major risk factors for an extraperitoneal anastomotic leak include: The distance of the anastomosis from the anal verge (Patients with a low anterior resection and an anastomosis within 5 cm from the anal verge are the highest risk group for an anastomotic leak), Anastomotic ischemia, Male gender, Obesity.

Major risk factors for an intraperitoneal anastomotic leak include: American Society of Anesthesiologists (ASA) score Grade III to V, Emergent surgery, Prolonged operative time, Handsewn ileocolic anastomosis.

Controversial, inconclusive, or pertinent negative associations between the following variables and an anastomotic leak have been reported: Neoadjuvant radiation therapy, Drains, Protective stoma, Hand-sewn colorectal anastomosis, Laparoscopic procedure, Mechanical bowel preparation, Nutritional status, Perioperative corticosteroids.

Early diagnosis is crucial to treat patients limiting the related mortality. For this reason several clinical items were proposed in literature to detect anastomotic leakage as soon as possible: fever, pain, tachycardia, peritoneal, purulent or faecal drain, and dynamic ileus [1-5]. Moreover, also laboratory markers were proposed, such as leukocytosis, serum procalcitonin (PCT) and C-Reactive Protein (CRP) [11-13]. Finally, in 2009 den Dulk et al. [14] proposed a leakage score (DUtch LeaKage, DULK), that consider several items (fever, heart rate, respiratory rate, urinary production, mental status, clinical conditions, signs of ileus, gastric retention, fascial dehiscence, abdominal pain, wound pain, leukocytosis, CRP, increase of urea or creatinine and nutrition status), to give a score, based on which is chosen a therapeutic strategy.

Therefore, we planned this study to prospectively evaluate anastomotic leakage rate after colorectal resections, trying to give a definite answer to the need for clear risk factors, and testing the diagnostic yeald of DULK score and laboratory markers.

#### **METHODS**

Prospective enrollment from September 2017 to November 2018 in 20 Italian surgical centers. All patients undergoing elective colorectal surgery with anastomosis will be included in a prospective database after having provided a written informed consent. A total of more than 1,160 patients is expected based on a mean of 50 cases/year per center.

# **Inclusion criteria**

- 1. Patients submitted to laparoscopic/open/converted ileo-colo-rectal resection with anastomosis (both intra- and extra-corporeal), including planned Hartmann's reversals.
- 2. American Society of Anesthesiologists' (ASA) class I, II or III
- 3. Elective surgery
- 4. Patients' written acceptance to be included in the study.

# **Exclusion criteria**

- 1. American Society of Anesthesiologists' (ASA) class IV-V
- 2. Patients with stoma before or at operation
- 3. Simple stoma closure
- 4. Transanal procedure
- 5. Pregnancy
- 6. Ongoing infection prior to surgery
- 7. Hyperthermic intraperitoneal chemotherapy for carcinomatosis.

# **Outcome measures**

 Preoperative risk factors of anastomotic leakage (age, gender, obesity, state of nutrition [9-10], diabetes, cardiovascular, renal failure, inflammatory bowel disease, ASA class I-II vs III)

- Operative parameters (approach, procedure, anastomotic technique, time of operation, pTNM stage)
- 3. Leukocyte count, serum CRP, serum procalcitonin and DULK score assessment in 2<sup>nd</sup> and 3<sup>rd</sup> postoperative day. Minor and major complications according to Clavien-Dindo classification [15, 16]
- 4. Anastomotic leakage rate
- 5. Morbidity-Mortality rates
- 6. Length of postoperative hospital stay

# Recorded data and follow-up

Potential patient-specific and intraoperative risk factors will be recorded: gender, body mass index, nutritional status according to the Mini Nutritional Assessment short-form [17, 18], surgical indication (cancer, polyps, chronic inflammatory bowel disease, diverticular disease), preoperative albuminemia, use of steroids, renal failure and dialysis, preoperative leukocyte count, CRP, PCT cardiovascular or respiratory disease, American Society of Anesthesia score, bowel preparation (decision made by operating surgeon), laparoscopy or laparotomy, level of anastomosis and technique (mechanical or hand-sewn, intra- or extra-corporeal), operative time, presence of drainage, surgeon and perioperative blood transfusion(s). During the postoperative period, patients will be examined by the attending surgeon daily. Fever (central temperature > 38 °C), pulse, abdominal signs, bowel movements, volume and aspect of drainage (if present) will be recorded daily. Leucocyte count, CRP, PCT and Dulk score will be measured in the evening before the operation (in addition to albuminemia) and on postoperative days 2, 3, and 6 (optional). The attending surgeon will make any decision for complementary exams and imaging according to his own criteria. The rate of any complication will be calculated and graded according to Clavien-ALL 3 – Protocollo dello Studio

Dindo [15, 16] including all leaks (independently of clinical significance), wound infection, pneumonia, central line infection, urinary tract infection. Urinary tract infection will be diagnosed on the basis of positive urine culture with bacterial count. Central line infection will be diagnosed on the basis of positive blood culture. Superficial and deep incisional infections will be diagnosed according to the definitions of the Centers for Disease Control and Prevention and a culture will be performed [19]. Pneumonia will be diagnosed on the basis of clinical symptoms, and physical and radiological examinations. The surgeons will be blinded to the results of the CRP and PCT assays. Patients will be followed-up in the outpatient clinic up to 6 weeks after discharge from the hospital.

Main outcome is anastomotic dehiscence (intended as any deviation from the planned postoperative course related to the anastomosis, or presence of pus or enteric contents within the drains, presence of abdominal or pelvic collection in the area of the anastomosis on postoperative CT scan, performed at the discretion of the attending surgeon, leakage of contrast through the anastomosis during enema or evident anastomotic dehiscence at reoperation for postoperative peritonitis). Thus, all detected leaks will be considered independently of clinical significance. No imaging will be performed routinely in order to search for leakage.

Secondary outcomes are morbidity and mortality rates, and postoperative length of stay. All data will be prospectively recorded into CRF and transmitted to the coordinating center on a monthly basis. Thereafter, all data will be incorporated into a spreadsheet (MS Excel), checking for any discrepancy, that will be addressed and solved through strict cooperation between chief investigator, data manager and participating center.

# **Statistical Analysis**

Quantitative values will be expressed as mean ± standard deviation, median and range; categorical data with percentage frequencies. Mean values of duration of stay will be compared according to the presence or absence of fistulas using Student's two-sided t test (allowing for heterogeneity of variances) or with a non-parametric Mann-Whitney test. Mean values of DULK score, CRP and PCT levels will also be compared using Student's two-sided t test (allowing for heterogeneity of variances) or with a non-parametric Mann-Whitney test. Both univariate analysis and multivariate analysis will be performed to assess risk factors for leakage and overall complications. The odds ratio (OR) will be presented followed by its 95% confidence interval (95% CI). Areas under the receiver-operating characteristics (ROC) curve will be calculated. For all statistical tests the significant level is fixed at p < .05. Multivariate analysis will be performed using logistic models. Statistical analyses will be carried out using STATA software (Stata Corp. College Station, Texas, USA).

# Sample size

Considering that the ASA grade (I and II vs. III) is mostly significant among risk factors for anastomotic dehiscence [3, 5, 8], an estimation of the OR for anastomotic dehiscence and ASA grade is equal to 5.6 [20]; assuming a confidence interval for the estimation of the OR at 95% and a maximum error equal to 0.04, the required sample size is n=1,062 (about 885 and 177 cases expected in ASA I-II and ASA III, respectively).

# REFERENCES

- Boushey R, Williams LJ. Management of anastomotic complications of colorectal surgery.
   Uptodate 2017.
- Slieker JC, Komen N, Mannaerts GH, et al. Long-term and perioperative corticosteroids in anastomotic leakage: a prospective study of 259 left-sided colorectal anastomoses. Arch Surg 2012; 147:447.
- 3. Kingham TP, Pachter HL. Colonic anastomotic leak: risk factors, diagnosis, and treatment. J Am Coll Surg 2009; 208:269.
- 4. Hyman N, Manchester TL, Osler T, et al. Anastomotic leaks after intestinal anastomosis: it's later than you think. Ann Surg 2007; 245:254-8.
- 5. Park JS, Choi GS, Kim SH, et al. Multicenter analysis of risk factors for anastomotic leakage after laparoscopic rectal cancer excision: the Korean laparoscopic colorectal surgery study group. Ann Surg 2013; 257:665.
- 6. Dietz, DW, Bailey, HR. Postoperative complications. In: ASCRS Textbook of Colon and Rectal Surgery, Church, JM, Beck, DE, Wolff, BG, Fleshman, JW, Pemberton, JH, (Eds), Springer-Verlag New York, LLC, New York 2006. p.141.
- 7. Bruce J, Krukowski ZH, Al-Khairy G, et al. Systematic review of the definition and measurement of anastomotic leak after gastrointestinal surgery. Br J Surg 2001; 88:1157.
- 8. Law WI, Chu KW, Ho JW, Chan CW. Risk factors for anastomotic leakage after low anterior resection with total mesorectal excision. Am J Surg 2000; 179:92.
- 9. Lipska MA, Bissett IP, Parry BR, Merrie AE. Anastomotic leakage after lower gastrointestinal anastomosis: men are at a higher risk. ANZ J Surg 2006; 76:579.
- 10. Platell C, Barwood N, Dorfmann G, Makin G. The incidence of anastomotic leaks in patients undergoing colorectal surgery. Colorectal Dis 2007; 9:71.
- 11. Giaccaglia V, Salvi PF, Cunsolo GV, Sparagna A, Antonelli MS, Nigri G, Balducci G, Ziparo V. Procalcitonin, as an early biomarker of colorectal anastomotic leak, facilitates enhanced recovery after surgery. J Crit Care 2014; 29:528-32.
- 12. Ortega-Deballon P, Radais F, Facy O, d'Athis P, Masson D, Charles PE, Cheynel N, Favre JP, Rat P. C-reactive protein is an early predictor of septic complications after elective colorectal surgery. World J Surg 2010; 34:808-14.

- 13. Oberhofer D, Juras J, Pavicić AM, Rancić Zurić I, Rumenjak V. Comparison of C-reactive protein and procalcitonin as predictors of postoperative infectious complications after elective colorectal surgery. Croat Med J 2012; 53:612-9.
- 14. den Dulk M, Noter SL, Hendriks ER, Brouwers MA, van der Vlies CH, Oostenbroek RJ, Menon AG, Steup WH, van de Velde CJ. Improved diagnosis and treatment of anastomotic leakage after colorectal surgery. Eur J Surg Oncol 2009; 35:420-6.
- 15. Dindo D, Demartines N, Clavien PA. Classification of surgical complications. A new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg 2004; 240:205-13.
- 16. Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibañes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. (2009). The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg Aug;250(2):187-96.
- 17. Kaiser MJ, Bauer JM, Ramsch C, Uter W, Guigoz Y, Cederholm T, Thomas DR, Anthony P, Charlton KE, Maggio M, Tsai AC, Grathwohl D, Vellas B, Sieber CC, MNA-International Group. Validation of the Mini Nutritional Assessment short-form (MNA-SF): a practical tool for identification of nutritional status. J Nutr Health Aging. 2009;13(9):782.
- 18. Skipper A, Ferguson M, Thompson K, Castellanos VH, Porcari J. Nutrition screening tools: an analysis of the evidence. JPEN J Parenter Enteral Nutr 2012; 36:292-8.
- 19. Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG. CDC definitions of nosocomial surgical site infections 1992: a modification of CDC definitions of surgical wound infections. Infect Control Hosp Epidemiol. 1992;13:606–8.
- 20. Choi HK, Law WL, Ho JWC. Leakage after resection and intraperitoneal anastomosis for colorectal malignancy: analysis of risk factors. Dis Colon Rectum 2006; 49:1719-1725

# Appendix 1 DULK SCORE [14]

| | Valori Normali | Score | Valori alterati | Score |
|---|---|---|---|---|
| Febbre | ≤ 38.0° C | 0 | ≥ 38.0° C | 1 |
| Frequenza cardiaca | ≤ 100 bpm | 0 | ≥ 100 bpm | 1 |
| Frequenza respiratoria | ≤ 30 atti/min | 0 | ≥ 30 atti/min | 1 |
| Diuresi | ≥ 30 ml/h o 700 ml/die | 0 | ≤ 30 ml/h o 700 ml/die | 1 |
| Stato mentale | Normale stato mentale | 0 | Agitazione o Letargia | 2 |
| Condizioni cliniche | Stabili o in miglioramento | 0 | Deterioramento | 2 |
| Segni di ileo | No | 0 | Ileo | 2 |
| Ritenzione gastrica | No | 0 | Ritenzione Gastrica | 2 |
| Deiscenza della fascia | No | 0 | Deiscenza della fascia | 2 |
| Dolore addominale o altri non di ferita | No dolore | 0 | Dolore non della ferita | 2 |
| Segni di infezione | No aumento leucociti o PCR | 0 | Aumento dei leucociti<br>di ≥ 5% o della PCR | 1 |
| Funzionalità renale | No aumento Urea o<br>Creatinina | 0 | Aumento di Urea o<br>Creatinina di ≥ 5% | 1 |
| Stato nutrizionale | Dieta Normale | 0 | Enterale/Parenterale Totale | 1/2 |
| TOTALE | | | | |

# Appendix 2 CLAVIEN-DINDO CLASSIFICATION [15, 16]

**TABLE 1.** Classification of Surgical Complications

#### **Grade Definition**

Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions

Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics, electrolytes, and physiotherapy. This grade also includes wound infections opened at the bedside

Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications

Blood transfusions and total parenteral nutrition are also included

Grade III Requiring surgical, endoscopic or radiological intervention

Grade IIIa Intervention not under general anesthesia

Grade IIIb Intervention under general anesthesia

Grade IV Life-threatening complication (including CNS complications)\* requiring IC/ICU management

Grade IVa Single organ dysfunction (including dialysis)

Grade IVb Multiorgan dysfunction

Grade V Death of a patient

Suffix "d" If the patient suffers from a complication at the time of discharge (see examples in Table 2), the suffix "d" (for "disability") is added to the respective grade of complication. This label indicates the need for a follow-up to fully evaluate the complication.

\*Brain hemorrhage, ischemic stroke, subarrachnoidal bleeding, but excluding transient ischemic attacks.

CNS, central nervous system; IC, intermediate care; ICU, intensive care unit.

**TABLE 2.** Clinical Examples of Complication Grades

| Grade I Respiratory Neurological Gastrointestinal Renal Transient confusion not requiring therapy Neurological Gastrointestinal Renal Transient clevation of serum creatinine Other Wound infection treated by opening of the wound at the bedside Grade II Grade II Grade II Grade II Grade III Gra | Grades | Organ System | Examples |
|---|---|---|---|
| Neurological Gastrointestinal Renal Transient confusion not requiring therapy | Grade I | Cardiac | Atrial fibrillation converting after correction of Klevel |
| Gastrointestinal Renal Renal Transient elevation of serum creatinine Other Wound infection treated by opening of the wound at the bedside Grade II Gradiac Respiratory Neurological Renal Gastrointestinal Renal Urinary tract infection requiring antibiotics Other Grade IIIa Grade II | | Respiratory | |
| Grade II Renal Other Wound infection treated by opening of the wound at the bedside Grade II Cardiac Tachyarrhythmia requiringreceptor antagonists for heart rate control Respiratory Pneumonia treated with antibiotics on the ward TIA requiring treatment with anticoagulants Gastrointestinal Renal Urinary tract infection requiring antibiotics Other Same for I followed by tx with antibiotics for phlegmonous infection Grade IIIa Gradiac Bradyarrhythmia requiring pacemaker implantation in local anesthesia See grade IV Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by stenting Other Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac Cardiac temponade after thoracic surgery requiring fenestration Respiratory Neurological See grade IV Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by stenting Other Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac temponade after thoracic surgery requiring fenestration Respiratory Bronchopleural fistulas after thoracic surgery requiring surgical closure See grade IV Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by surgery Other Wound infection leading to eventration of small bowel Grade IVa Cardiac Heart failure leading to low-output syndrome Lung failure requiring intubation Neurological Ischemic stroke/brain hemorrhage Gastrointestinal Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Same as for IVa but in combination with renal failure Gastrointestinal Same as for IVa but in combination with hemodynamic instability Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | Neurological | Transient confusion not requiring therapy |
| Grade II Other Wound infection treated by opening of the wound at the bedside Cardiac Tachyarrhythmia requiringreceptor antagonists for heart rate control Pneumonia treated with antibiotics on the ward TIA requiring treatment with anticoagulants Infectious diarrhea requiring antibiotics Renal Urinary tract infection requiring antibiotics Other Same for I followed by tx with antibiotics for phlegmonous infection Grade IIIa Cardiac Bradyarrhythmia requiring pacemaker implantation in local anesthesia Neurological See grade IV Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by stenting Other Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac Emponade after thoracic surgery requiring surgical closure Neurological See grade IV Gastrointestinal Respiratory Neurological Stenosis of the ureter after kidney transplantation treated by stenting Other Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac temponade after thoracic surgery requiring fenestration Respiratory See grade IV Gastrointestinal Anastomotic leakage after descendorectostomy requiring relaparotomy Renal Stenosis of the ureter after kidney transplantation treated by surgery Other Wound infection leading to eventration of small bowel Grade IVa Cardiac Heart failure leading to low-output syndrome Respiratory Lung failure requiring intubation Neurological Ischemic stroke/brain hemorrhage Gastrointestinal Renal insufficiency requiring dialysis Grade IVb Cardiac Same as for IVa but in combination with renal failure Gastrointestinal Same as for IVa but in combination with hemodynamic instability Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | Gastrointestinal | Noninfectious diarrhea |
| Grade II Cardiac Respiratory Neurological Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by stenting Respiratory Neurological Gastrointestinal Renal User Grade IVb Cardiac Respiratory Neurological Renal Same as for IVa but in combination with renal failure Gastrointestinal Renal Respiratory Gastrointestinal Respiratory Gastrointestinal Respiratory Gastrointestinal Respiratory Gastrointestinal Respiratory Gastrointestinal Respiratory Neurological Gastrointestinal Respiratory Neurological See grade IV Stenosis of the ureter after kidney transplantation treated by surgery Stenosis of the ureter after kidney transplantation treated by surgery Stenosis of the ureter after kidney transplantation treated by surgery Stenosis of the ureter after kidney transplantation treated by surgery Other Wound infection leading to eventration of small bowel Cardiac Heart failure leading to low-output syndrome Lung failure requiring intubation Neurological Same as for IVa but in combination with renal failure Same as for IVa but in combination with remodynamic instability Ischemic stroke/brain hemorrhage with respiratory failure | | Renal | Transient elevation of serum creatinine |
| Respiratory Neurological Gastrointestinal Renal Other Grade IIIa Gastrointestinal Renal Other Grade IIIa Gastrointestinal Renal Other Grade IIIa Gastrointestinal Renal Other Grade IIIa Gastrointestinal Renal Neurological Renal Other Gastrointestinal Renal Other Gastrointestinal Renal Other Grade IIIb Gastrointestinal Renal Other Grade IIIb Gastrointestinal Renal Other Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac temponade after thoracic surgery requiring fenestration Respiratory Neurological Renal Renal Stenosis of the ureter after kidney transplantation treated by stenting Other Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac temponade after thoracic surgery requiring fenestration Respiratory Neurological Renal Renal Stenosis of the ureter after kidney transplantation treated by surgery Other Wound infection leading to eventration of small bowel Grade IVa Respiratory Neurological Gastrointestinal Renal Gastrointestinal Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Respiratory Same as for IVa but in combination with renal failure Gastrointestinal Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | Other | Wound infection treated by opening of the wound at the bedside |
| Neurological Gastrointestinal Renal Urinary tract infectious diarrhea requiring antibiotics Other Same for I followed by tx with antibiotics for phlegmonous infection Bradyarrhythmia requiring pacemaker implantation in local anesthesia Neurological Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by stenting Other Closure of dehiscent noninfected wound in the OR under local anesthesia Grade IIIb Cardiac Cardiac temponade after thoracic surgery requiring surgical closure See grade IV Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by stenting Other Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac temponade after thoracic surgery requiring fenestration Bronchopleural fistulas after thoracic surgery requiring surgical closure See grade IV Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by surgery Other Wound infection leading to eventration of small bowel Grade IVa Cardiac Heart failure leading to low-output syndrome Respiratory Neurological Gastrointestinal Renal Renal insufficiency requiring intubation Grade IVb Cardiac Same as for IVa but in combination with renal failure Gastrointestinal Neurological Ischemic stroke/brain hemorrhage with respiratory failure Same as for IVa but in combination with renal failure Same as for IVa but in combination with respiratory failure | Grade II | Cardiac | Tachyarrhythmia requiringreceptor antagonists for heart rate control |
| Gastrointestinal Renal Urinary tract infection requiring antibiotics Other Same for I followed by tx with antibiotics for phlegmonous infection Grade IIIa Cardiac Bradyarrhythmia requiring pacemaker implantation in local anesthesia Neurological See grade IV Gastrointestinal Biloma after liver resection requiring percutaneous drainage Renal Stenosis of the ureter after kidney transplantation treated by stenting Other Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac Cardiac temponade after thoracic surgery requiring fenestration Respiratory Bronchopleural fistulas after thoracic surgery requiring surgical closure Neurological See grade IV Gastrointestinal Anastomotic leakage after descendorectostomy requiring relaparotomy Stenosis of the ureter after kidney transplantation treated by surgery Other Wound infection leading to eventration of small bowel Grade IVa Cardiac Heart failure leading to low-output syndrome Respiratory Lung failure requiring intubation Neurological Ischemic stroke/brain hemorrhage Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Same as for IVa but in combination with renal failure Respiratory Same as for IVa but in combination with hemodynamic instability Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | Respiratory | Pneumonia treated with antibiotics on the ward |
| Renal Urinary tract infection requiring antibiotics Other Same for I followed by tx with antibiotics for phlegmonous infection Grade IIIa Cardiac Bradyarrhythmia requiring pacemaker implantation in local anesthesia Neurological See grade IV Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by stenting Other Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac Cardiac temponade after thoracic surgery requiring fenestration Respiratory Bronchopleural fistulas after thoracic surgery requiring surgical closure See grade IV Gastrointestinal Anastomotic leakage after descendorectostomy requiring relaparotomy Renal Stenosis of the ureter after kidney transplantation treated by surgery Other Wound infection leading to eventration of small bowel Grade IVa Cardiac Heart failure leading to low-output syndrome Respiratory Neurological Ischemic stroke/brain hemorrhage Gastrointestinal Renal Renal Insufficiency requiring dialysis Grade IVb Cardiac Same as for IVa but in combination with renal failure Respiratory Same as for IVa but in combination with hemodynamic instability Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | Neurological | TIA requiring treatment with anticoagulants |
| Grade IIIa Other Cardiac Reurological Renal Other Cardiac Respiratory Other Other Castrointestinal Renal Gastrointestinal Respiratory Other Castrointestinal Renal Cardiac Gastrointestinal Respiratory Neurological Gastrointestinal Renal Cardiac Cardiac the ureter after kidney transplantation treated by stenting Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac temponade after thoracic surgery requiring fenestration Bronchopleural fistulas after thoracic surgery requiring surgical closure See grade IV Anastomotic leakage after descendorectostomy requiring relaparotomy Renal Stenosis of the ureter after kidney transplantation treated by surgery Other Wound infection leading to eventration of small bowel Cardiac Heart failure leading to low-output syndrome Lung failure requiring intubation Neurological Gastrointestinal Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Same as for IVa but in combination with renal failure Respiratory Same as for IVa but in combination with hemodynamic instability Ischemic stroke/brain hemorrhage with respiratory failure | | Gastrointestinal | Infectious diarrhea requiring antibiotics |
| Grade IIIa Cardiac Neurological See grade IV Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by stenting Other Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac Earlie IV Bronchopleural fistulas after thoracic surgery requiring fenestration Respiratory Neurological Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by stenting Other Cardiac temponade after thoracic surgery requiring fenestration Respiratory Bronchopleural fistulas after thoracic surgery requiring surgical closure See grade IV Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by surgery Other Wound infection leading to eventration of small bowel Grade IVa Cardiac Heart failure leading to low-output syndrome Lung failure requiring intubation Neurological Ischemic stroke/brain hemorrhage Gastrointestinal Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Same as for IVa but in combination with renal failure Respiratory Same as for IVa but in combination with renal failure Same as for IVa but in combination with hemodynamic instability Ischemic stroke/brain hemorrhage with respiratory failure | | Renal | Urinary tract infection requiring antibiotics |
| Neurological Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by stenting Other Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac Earlier Earl | | Other | Same for I followed by tx with antibiotics for phlegmonous infection |
| Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by stenting Other Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac Cardiac temponade after thoracic surgery requiring fenestration Respiratory Neurological See grade IV Gastrointestinal Renal Other | Grade IIIa | Cardiac | Bradyarrhythmia requiring pacemaker implantation in local anesthesia |
| Renal Other Closure of dehiscent noninfected wound in the OR under local anesthesia Cardiac Cardiac temponade after thoracic surgery requiring fenestration Respiratory Neurological See grade IV Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by surgery other Wound infection leading to eventration of small bowel Grade IVa Cardiac Heart failure leading to low-output syndrome Respiratory Neurological Ischemic stroke/brain hemorrhage Gastrointestinal Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Same as for IVa but in combination with renal failure Respiratory Same as for IVa but in combination with hemodynamic instability Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | Neurological | See grade IV |
| Grade IIIb Cardiac Cardiac temponade after thoracic surgery requiring fenestration Respiratory Neurological Renal Cardiac Eastrointestinal Renal Respiratory Other Wound infection leading to eventration of small bowel Grade IVa Respiratory Neurological Gastrointestinal Respiratory Other Grade IVa Respiratory Neurological Respiratory Neurological Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by surgery Other Wound infection leading to eventration of small bowel Cardiac Heart failure leading to low-output syndrome Respiratory Neurological Gastrointestinal Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Respiratory Gastrointestinal Neurological Same as for IVa but in combination with renal failure Respiratory Gastrointestinal Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | Gastrointestinal | Biloma after liver resection requiring percutaneous drainage |
| Grade IIIb Cardiac Respiratory Neurological Renal Grade IV Grade | | Renal | Stenosis of the ureter after kidney transplantation treated by stenting |
| Respiratory Neurological See grade IV Gastrointestinal Renal Grade IVa Gastrointestinal Respiratory Other Respiratory Other Respiratory Other Respiratory Remal Respiratory Neurological Gastrointestinal Renal Gastrointestinal Renal Gastrointestinal Renal Respiratory Neurological Gastrointestinal Renal Respiratory Gastrointestinal Renal Respiratory Gastrointestinal Renal Respiratory Gastrointestinal Respiratory Gastrointestinal Respiratory Gastrointestinal Respiratory Gastrointestinal Neurological Gastrointestinal Neurological Gastrointestinal Neurological Same as for IVa but in combination with renal failure Gastrointestinal Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | Other | Closure of dehiscent noninfected wound in the OR under local anesthesia |
| Neurological Gastrointestinal Renal Other Wound infection leading to eventration of small bowel Grade IVa Respiratory Neurological Gastrointestinal Renal Gastrointestinal Renal Gastrointestinal Renal Respiratory Neurological Gastrointestinal Renal Respiratory Same as for IVa but in combination with renal failure Gastrointestinal Neurological Gastrointestinal Respiratory Gastrointestinal Respiratory Gastrointestinal Neurological Gastrointestinal Neurological Gastrointestinal Neurological Same as for IVa but in combination with renal failure Same as for IVa but in combination with hemodynamic instability Neurological Ischemic stroke/brain hemorrhage with respiratory failure | Grade IIIb | | |
| Gastrointestinal Renal Stenosis of the ureter after kidney transplantation treated by surgery Other Wound infection leading to eventration of small bowel Cardiac Heart failure leading to low-output syndrome Respiratory Neurological Gastrointestinal Renal Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Respiratory Gastrointestinal Respiratory Gastrointestinal Respiratory Gastrointestinal Neurological Same as for IVa but in combination with renal failure Same as for IVa but in combination with hemodynamic instability Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | Respiratory | Bronchopleural fistulas after thoracic surgery requiring surgical closure |
| Renal Stenosis of the ureter after kidney transplantation treated by surgery Other Wound infection leading to eventration of small bowel Grade IVa Cardiac Heart failure leading to low-output syndrome Respiratory Lung failure requiring intubation Neurological Ischemic stroke/brain hemorrhage Gastrointestinal Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Same as for IVa but in combination with renal failure Respiratory Gastrointestinal Neurological Ischemic stroke/brain hemorrhage with respiratory failure Ischemic stroke/brain hemorrhage with respiratory failure | | Neurological | See grade IV |
| Other Wound infection leading to eventration of small bowel Grade IVa Cardiac Heart failure leading to low-output syndrome Respiratory Lung failure requiring intubation Neurological Ischemic stroke/brain hemorrhage Gastrointestinal Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Same as for IVa but in combination with renal failure Respiratory Gastrointestinal Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | Gastrointestinal | |
| Grade IVa Respiratory Neurological Gastrointestinal Renal Grade IVb Cardiac Respiratory Necrotizing pancreatitis Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Respiratory Gastrointestinal Neurological Neurological Same as for IVa but in combination with renal failure Respiratory Gastrointestinal Neurological Same as for IVa but in combination with hemodynamic instability Ischemic stroke/brain hemorrhage with respiratory failure | | Renal | |
| Respiratory Lung failure requiring intubation Neurological Ischemic stroke/brain hemorrhage Gastrointestinal Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Same as for IVa but in combination with renal failure Respiratory Gastrointestinal Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | | |
| Neurological Gastrointestinal Renal Ischemic stroke/brain hemorrhage Grade IVb Cardiac Same as for IVa but in combination with renal failure Respiratory Gastrointestinal Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | | |
| Gastrointestinal Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Respiratory Gastrointestinal Neurological Necrotizing pancreatitis Renal insufficiency requiring dialysis Same as for IVa but in combination with renal failure Same as for IVa but in combination with renal failure Same as for IVa but in combination with hemodynamic instability Ischemic stroke/brain hemorrhage with respiratory failure | | | |
| Renal Renal insufficiency requiring dialysis Grade IVb Cardiac Same as for IVa but in combination with renal failure Respiratory Same as for IVa but in combination with renal failure Gastrointestinal Same as for IVa but in combination with hemodynamic instability Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | | |
| Grade IVb Cardiac Same as for IVa but in combination with renal failure Respiratory Same as for IVa but in combination with renal failure Gastrointestinal Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | | |
| Respiratory Same as for IVa but in combination with renal failure Gastrointestinal Same as for IVa but in combination with hemodynamic instability Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | | |
| Gastrointestinal Same as for IVa but in combination with hemodynamic instability Neurological Ischemic stroke/brain hemorrhage with respiratory failure | Grade IVb | | |
| Neurological Ischemic stroke/brain hemorrhage with respiratory failure | | 1 2 | |
| Renal Same as for IVa but in combination with hemodynamic instability | | | |
| Suffix "d" Cardia Cardia insufficiency of the my coordial inferentian (No. d) | | Renal | Same as for IVa but in combination with hemodynamic instability |

Suffix "d" Cardiac Cardiac insufficiency after myocardial infarction (IVa-d)

Respiratory Dyspnea after pneumonectomy for severe bleeding after chest tube placement (IIIb-d)

Gastrointestinal Residual fecal incontinence after abscess following descendorectostomy with surgical evacuation. (IIIb-d)

Neurological Stroke with sensorimotor hemisyndrome (IVa-d)

Renal Residual renal insufficiency after sepsis with multiorgan dysfunction (IVb-d)

Other Hoarseness after thyroid surgery (I–d) TIA, transient ischemic attack; OR, operating room.

# Appendix 3 MNA® [17]

# **Screening**

```
A Presenta una perdita dell' appetito? Ha mangiato meno negli ultimi 3 mesi? (perdita d'appetito,
   problemi digestivi, difficoltà di masticazione o deglutizione)
   0 = Grave riduzione dell'assunzione di cibo
   1 = Moderata riduzione dell'assunzione di cibo
   2 = Nessuna riduzione dell'assunzione di cibo
B Perdita di peso recente (<3 mesi)
   0 = perdita di peso > 3 kg
   1 = non sa
   2 = perdita di peso tra 1 e 3 kg
   3 = nessuna perdita di peso
C Motricità
   0 = dal letto alla poltrona
   1 = autonomo a domicilio
   2 = esce di casa
D Nell' arco degli ultimi 3 mesi: malattie acute o stress psicologici?
   0 = si 2 = no
E Problemi neuropsicologici
```

0 = demenza o depressione grave

1 = demenza moderata

2 = nessun problema psicologico

# F1 Indice di massa corporea (IMC) = peso in kg / (alt ezza in m)

0 = IMC < 191 = 19 ≤ IMC < 21  $2 = 21 \le IMC < 23$ 3 = IMC ≥ 23

SE L'IMC NON E DISPONIBILE, SOSTITUIRE LA DOMANDA F1 CON LA DOMANDA F2.

NON RISPONDERE ALLA DOMANDA F2 SE LA DOMANDA F1 E GIA' STATA COMPLETATA

#### F2 Circonferenza del polpaccio (CP in cm)

0 = CP inferiore a 31 3 = CP 31 o superiore

# Valutazione di screening (max.14 punti)

12-14 punti: stato nutrizionale normale 8-11 punti: a rischio di malnutrizione

0-7 punti: malnutrito

Ref. Vellas B, Villars H, Abellan G, et al. Overview of the MNA® - Its History and Challenges. J Nutr Health Aging 2006;10:456-465.

Rubenstein LZ, Harker JO, Salva A, Guigoz Y, Vellas B. Screening for Undernutrition in Geriatric Practice: Developing the Short-Form Mini Nutritional Assessment (MNA-SF). J. Geront 2001;56A: M366-377.

Guigoz Y. The Mini-Nutritional Assessment (MNA®) Review of the Literature - What does it tell us? J Nutr Health Aging 2006; 10:466-487. Kaiser MJ, Bauer JM, Ramsch C, et al. Validation of the Mini Nutritional Assessment Short-Form (MNA®-SF): A practical tool for identification of nutritional status. J Nutr Health Aging 2009; 13:782-788.

® Société des Produits Nestlé, S.A., Vevey, Switzerland, Trademark Owners

© Nestlé, 1994, Revision 2009. N67200 12/99 10M

Per maggiori informazioni: www.mna-elderly.com

# Appendix 4

<u>Chief Investigator</u>: Marco Catarci, MD – UOC Chirurgia Generale – Ospedale Mazzoni – Via degli

Iris snc; 63100 Ascoli Piceno – AV 5 – ASUR Marche – email: <a href="mailto:marcocatarci@gmail.com">marcocatarci@gmail.com</a>;

marco.catarci@sanita.marche.it; cellulare: 329-8610040.

Statistical Advisor & Data Manager: Benedetta Ruggeri, MD, PhD - UOS Governo Clinico - AV 5 -

Via degli Iris snc; 63100 Ascoli Piceno –ASUR Marche – email: <a href="mailto:benedetta.ruggeri@sanita.marche.it">benedetta.ruggeri@sanita.marche.it</a>;